CLINICAL TRIAL: NCT00096785
Title: Randomized, Open-Label, Comparative Study to Evaluate Early Viral Load Reductions and Exploratory Viral Kinetics Following Administration of Entecavir or Adefovir in Nucleoside-Naive Adults With Chronic Hepatitis B Infection
Brief Title: Comparative Trial of Entecavir Versus Adefovir in the Treatment of Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-079
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-06

CONDITIONS: Hepatitis B; Chronic Disease
Keywords: chronic hepatitis B infection
MeSH Terms: conditions — Hepatitis B; Chronic Disease; Hepatitis B, Chronic | interventions — entecavir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: entecavir
- A2 (Active Comparator)
  Interventions: Drug: adefovir

INTERVENTIONS:
Drug: entecavir — Tablets, Oral, ETV 0.5 mg, once daily, up to 96 weeks
  Other Names: Baraclude
  Arms: A1
Drug: adefovir — Tablets, Oral, ADV 10 mg, once daily, up to 96 weeks
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate antiviral activity and efficacy of entecavir (ETV) compared to adefovir in adults with chronic hepatitis B who have not been treated yet with an antiviral medicine.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B treatment naive
* Compensated liver disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (11):
  - Local Institution, San Diego, California
  - Local Institution, San Francisco, California
  - Local Institution, Torrance, California
  - Local Institution, Miami, Florida
  - Local Institution, North Miami Beach, Florida
  - Local Institution, Baltimore, Maryland
  - Local Insitution, New York, New York
  - Local Institution, New York, New York
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Dallas, Texas
  - Local Institution, Galveston, Texas
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
- Hong Kong (3):
  - Local Institution, Chai Wan
  - Local Institution, Pokfulham
  - Local Institution, Tai Po
- Local Institution, Jakarta, Indonesia
- Philippines (2):
  - Local Institution, Cebu
  - Local Institution, Manila
- Local Institution, Singapore, Singapore
- Taiwan (2):
  - Local Institution, Taichung
  - Local Institution, Taoyan
- Local Institution, Bangkok, Thailand

REFERENCES:
- [Background] Leung N, Peng CY, Hann HW, Sollano J, Lao-Tan J, Hsu CW, Lesmana L, Yuen MF, Jeffers L, Sherman M, Min A, Mencarini K, Diva U, Cross A, Wilber R, Lopez-Talavera J. Early hepatitis B virus DNA reduction in hepatitis B e antigen-positive patients with chronic hepatitis B: A randomized international study of entecavir versus adefovir. Hepatology. 2009 Jan;49(1):72-9. doi: 10.1002/hep.22658. PMID 19065670

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 132 enrolled; 63 not randomized (59 did not meet study criteria, 3 withdrew consent, 1 lost to follow-up). 1 randomized to adefovir (ADV) received entecavir (ETV) throughout treatment, & is counted in the ADV group for primary efficacy analysis, not included in the secondary efficacy analyses, & counted in the ETV group in safety analyses.
Groups:
- Entecavir: ETV 0.5 mg once daily (QD)
- Adefovir: ADV 10 mg QD
Period: Overall Study
Arm/Group | Entecavir | Adefovir
Started | 35 (1 participant randomized to ADV, treated with ETV. (As randomized= 35; as treated=36)) | 34 (1 participant randomized to ADV, treated with ETV. (As randomized= 34; as treated=33))
As-Randomized Population | 35 | 34
As-Treated Population | 36 | 33
Completed | 33 (As randomized cohort) | 33 (As randomized cohort)
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Relocated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir | Adefovir | Total
Number analyzed (Participants) | 35 | 34 | 69
Age Continuous [Mean (Standard Deviation); unit: years] | 37 (2.3) | 32 (1.9) | 34 (1.5)
Age Continuous [Median (Full Range); unit: participants] | 38 [18 to 76] | 28 [17 to 57] | 31 [17 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 22 | 23 | 45
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 31 | 30 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  North America | 9 | 13 | 22
  East Asia | 26 | 21 | 47
Prior interferon (IFN) [Number; unit: Participants]
  Prior IFN | 1 | 1 | 2
  No prior IFN | 34 | 33 | 67
Alanine Aminotransferease (ALT) [Mean (Standard Deviation); unit: U/L] | 109.4 (81.76) | 176.4 (207.22) | 142.4 (159.12)
Hepatitis B virus DNA (HBV DNA) by Polymerase Chain Reaction (PCR) [Mean (Standard Deviation); unit: log10 copies/mL] | 10.45 (2.125) | 9.89 (1.201) | 10.18 (1.742)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatitis B Virus DNA (HBV DNA) by Polymerase Chain Reaction (PCR) Assay at Week 12
Description: Antiviral efficacy, as measured by the mean reduction in serum HBV DNA levels by PCR (log10 copies/mL) at Week 12, adjusted for baseline (Week 12 - baseline). A negative value = improvement.
Time Frame: Baseline, Week 12
Population: As-randomized participants who completed 12 weeks of treatment
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 33
log10 copies/mL | -6.23 (0.247) | -4.52 (0.357)

2. Secondary Outcome: Change From Baseline in HBV DNA by PCR Assay at Week 48
Description: Antiviral efficacy, as measured by the mean reduction in serum HBV DNA levels by PCR (log10 copies/mL) at Week 48, adjusted for baseline (Week 48 - Baseline). A negative value = improvement.
Time Frame: Baseline, Week 48
Population: Treated subjects who had both baseline and Week 12 HBV DNA measurements and who received the randomized treatment. 1 participant randomized to ADV actually received ETV and is not counted in secondary efficacy analyses.
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
log10 c/mL | -7.28 (0.327) | -5.08 (0.455)

3. Secondary Outcome: Viral Load Undetectable (HBV DNA <300 Copies/mL)
Description: Number of Subjects with HBV DNA <300 copies/mL by Roche COBAS® Amplicor (limit of quantitation 300 copies/mL)
Time Frame: Week 48
Population: Treated participants who had both baseline and Week 12 HBV DNA measurements and who received the randomized treatment. 1 participant randomized to ADV actually received ETV and is not counted in secondary efficacy analyses.
Measure: Number; unit: Participants
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
Participants | 19 | 6

4. Secondary Outcome: Alanine Aminotransferase (ALT) Normalization
Description: Number of participants with ALT ≤ 1 x upper limit of normal (ULN)
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
participants | 25 | 20

5. Secondary Outcome: HBV DNA Viral Kinetics Estimates of Exponential Decay Model - Efficacy in Blocking Virus Production and de Novo Infections
Description: The biphasic decline of HBV DNA is characterized via a 4-parameter exponential decay model previously published for HBV compounds. The model parameters of interest are the effectiveness of the drug in blocking virus production from infected cells (efficacy, ε) and effectiveness of the study treatment in blocking de novo infection of susceptible cells (η). The model parameters reflect the biphasic pattern that is typically observed after initiation of antiviral therapy. Parameters were estimated for each subject separately and then averaged within each treatment group.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percent effective
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
percent effective
  Efficacy in blocking virus production - ε | 99.87 | 99.46
  Effectiveness in blocking de novo infections - η | 6.07 | 5.87

6. Secondary Outcome: HBV DNA Viral Kinetics Estimates of Exponential Decay Model - Viral Clearance Rate and Infected Cell Death Rate
Description: The biphasic decline of HBV DNA is characterized via a 4-parameter exponential decay model previously published for HBV compounds. The model parameters of interest are the clearance rate of the free virus (c), the death rate of productively infected cells (δ), The model parameters reflect the biphasic pattern that is typically observed after initiation of antiviral therapy. Parameters were estimated for each subject separately and then averaged within each treatment group.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: per day
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
per day
  Viral Clearance - c | 1.70 | 0.91
  Infected cell death - δ | 0.08 | 0.04

7. Secondary Outcome: HBV DNA Viral Kinetics Estimates of Exponential Decay Model - Half-Life of Free Virus
Description: The biphasic decline of HBV DNA is characterized via a 4-parameter exponential decay model previously published for HBV compounds. An important derived parameter is the half-life of free virus (ie, the average amount of time for HBV particles in plasma to be reduced to half the initial level), calculated as 24*ln(2)/c. The model parameters reflect the biphasic pattern that is typically observed after initiation of antiviral therapy. Parameters were estimated for each subject separately and then averaged within each treatment group.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: hours
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
hours | 14.52 | 32.46

8. Secondary Outcome: HBV DNA Viral Kinetics - Spline Model
Description: This analysis uses a 3-parameter piece-wise linear model and describes the biphasic decline in HBV DNA (measured by PCR assay) through Week 12. The 3 parameters are the values for the 2 slopes, describing the first and second phase declines, respectively, and the estimated HBV DNA at the knot (at day 10; the time point where the 2 phases join). The biphasic viral decay kinetics for each treatment were obtained using a spline fitting procedure to estimate the 3 parameters for each subject; these estimates were then averaged within each treatment group.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: log10 copies/mL
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 33 | 32
log10 copies/mL
  First slope (first phase of viral decay) | -0.391 | -0.329
  Second slope (second phase of viral decay) | -0.034 | -0.024

9. Secondary Outcome: Summary of Safety - Most Frequent (> 10%) Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuations Due to AEs, and Deaths
Description: AE=new untoward medical occurrence or worsening of pre-existing medical condition regardless of causal relationship to treatment. SAE=untoward medical occurrence that is life-threatening, a congenital anomaly/birth defect, or an important medical event, or results in death, inpatient hospitalization/prolongation of hospitalization, or persistent/significant disability. AE grades: mild (1), moderate (2), severe (3), life-threatening (4), death (5). ALT flare= >2x baseline & >10x ULN up to end of therapy + 5 days. Hepatic SAE=SAEs consistent with worsening of hepatitis or hepatic decompensation.
Time Frame: cumulative through the end of on-treatment observation as available at the time of the Week 48 dataset
Population: As-treated population. 1 participant was randomized to ADV, but treated with ETV was counted in the ETV group.
Measure: Number; unit: Participants
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 36 | 33
Participants
  Death | 0 | 0
  Serious AE | 1 | 3
  Discontinuation due to AE | 0 | 1
  Malignant neoplasm | 0 | 0
  On Treatment: Any AE | 28 | 27
  On Treatment: Headache | 9 | 6
  On Treatment: Upper Respiratory Infection | 8 | 8
  On Treatment: Influenza | 6 | 4
  On Treatment: Nasopharyngitis | 4 | 6
  On Treatment: Pyrexia | 4 | 6
  On Treatment: Back Pain | 0 | 5
  On Treatment: Grade 3-4 AEs | 2 | 5
  ALT Flare | 0 | 1
  Hepatic SAE | 1 | 2

10. Secondary Outcome: Summary of Safety - Laboratory Abnormalities Reported as Clinical AEs
Description: Laboratory abnormalities reported as clinical AEs
Time Frame: Week 48
Population: As-treated population. 1 participant who was randomized to ADV, but treated with ETV was counted in the ETV group.
Measure: Number; unit: Participants
Arm/Group | Entecavir | Adefovir
Number analyzed (Participants) | 36 | 33
Participants
  ALT increased | 1 | 2
  Lipase increased | 1 | 2
  Blood phosphorus decreased | 0 | 1
  Liver function test abnormal | 0 | 1
  Platelet count decreased | 0 | 1
  Protein urine present | 0 | 1

ADVERSE EVENTS:
Arm/Group | ADV 10 mg | ETV 0.5 mg
Serious Adverse Events (participants affected / at risk) | 2/33 | 1/36
Other Adverse Events (participants affected / at risk) | 16/33 | 17/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADV 10 mg (N=33) | ETV 0.5 mg (N=36)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADV 10 mg (N=33) | ETV 0.5 mg (N=36)
LIPASE INCREASED (Investigations) | 2 | 0
HEADACHE (Nervous system disorders) | 5 | 8
DIZZINESS (Nervous system disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 2
INFLUENZA (Infections and infestations) | 2 | 4
NASOPHARYNGITIS (Infections and infestations) | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
MALAISE (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.